CLINICAL TRIAL: NCT03048760
Title: Magnetic Resonance Imaging (MRI) for the Delineation of Organs At Risk (OAR) and Target Volumes in Lung Cancer Patients
Acronym: MR-Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Elekta Limited (Industry)
Responsible Party: Principal Investigator, Sally Falk, Professor Corinne Favire-Finn, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17_RADIO_121
Record Dates: First submitted 2017-01-16; First posted 2017-02-09 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
Keywords: MRI scan; Organs at Risk
MeSH Terms: conditions — Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan (Experimental): All participants will undergo 2 MRI scans - 1 at the time of their radiotherapy planning scan & 1 after approx. 2 weeks of radiotherapy treatment.
  Interventions: Other: MRI scan

INTERVENTIONS:
Other: MRI scan — All participants will undergo 2 MRI scans - 1 at the time of their radiotherapy planning scans & 1 after approx. 2 weeks of radiotherapy treatment.

SUMMARY:
The Christie NHS Foundation Trust is one of seven sites worldwide within the Atlantic consortium that is developing the Elekta MR-Linac (MRL) prior to commercial release at the end of 2017. The MRL allows MR images of patients to be acquired before, during and following radiotherapy (RT). One area where The Christie is taking the lead within the consortium is the application of the MRL for lung imaging and treatment, an area where MRI has hardly been used.

MRI scans provide greater soft tissue contrast than CT scans which can aid in the accurate delineation of organs at risk (OAR) and tumour target volumes for MRL and routine treatment. In addition, MRI can provide real time imaging which can aid in the accurate motion characterisation of these volumes. The addition of functional diffusion weighted imaging (DWI) has also proven to be useful in the discrimination of malignant from benign lesions; for lymph node detection and for the differentiation of tumour from atelectasis.

Auto-contouring has the potential to speed workflows at various points in the clinical pathway. This may be inter-patient contour propagation used pre-treatment for plan creation, or may be during online or offline adaptive workflows propagating contours through imaging acquired as treatment progresses. In collaboration with industry the investigators will be testing such algorithms on these images retrospectively.

In addition, the investigators would also like to evaluate patients' experiences of CT and MRI scans and determine which scanning method is preferred. Other studies have explored patient experiences of MRI compared to CT but not in the lung cancer patient population.

DETAILED DESCRIPTION:
Participants on this study will have two MRI scans in addition to the CT treatment planning scan, which is standard of care and cone beam CT scans during treatment, which are also standard of care. One of the MR scans will be close to the start of treatment and the other will be approximately 2 weeks after the start of radiotherapy treatment. If the patient has had a PET scan within 4 weeks of the 1st MR scan then the PET images will also be used for target volume delineation. If the PET scan > 4 weeks old, it can be repeated as per standard practice.

The MRI protocol includes up to 60 minutes of scanning which will include anatomical, respiratory dynamic and functional diffusion weighted imaging (DWI). The patient will be set up according to the treatment position on the MR scanner, using flat couch. The MR scans will not be used for clinical decision making.

Clinicians will then contour organs at risk (OARs) and target volumes on both the CT (guided by PET if available) and MRI scans and contours will be compared to determine the usefulness of MRI for radiotherapy treatment planning.

The contoured data sets will be fully anonymised, and used in house and shared with Elekta to assist with the development of automatic contouring / tumour tracking software, comparing CT to cone beam CT (CBCT) tracking (standard of care) with MR to MR tracking (experimental).

To assess experiences of MRI and CT, participants will be asked to complete baseline self-report questionnaires and additional questionnaires after MRI and CT scans. A small sample of participants will also be invited to participate in a semi-structured interview to explore their experiences in greater depth.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III Non-Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer (SCLC) (histological diagnosis not mandatory)
* Tumour Characteristics:

  * Size ≥ 3 cm in diameter
  * Positions: range of tumour positions with at least 10 of the participants having lower lobe tumours
* Patients planned for radical radiotherapy
* Eastern Co-operative Oncology Group (ECOG) Performance Status (PS) 0-2

Exclusion Criteria:

* Any contraindications to MR identified after MR safety screening including completion of an MR Safety Screening Form
* Unable to lie supine for 60 minutes
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Measure differences between target and OAR volumes contoured on PET, CT and MRI images. | 18 months

SECONDARY OUTCOMES:
Measure differences in inter-patient OAR volumes and intra-patient target and OAR volumes using MRI and CT. | 18 months
Measure patient experiences of CT and MRI using questionnaires and interviews. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, PhD, Principal Investigator — University of Manchester & The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The contoured data sets will be fully anonymised, and used in house and shared with Elekta to assist with the development of automatic contouring / tumour tracking software, comparing CT to cone beam CT (CBCT) tracking (standard of care) with MR to MR tracking (experimental).